CLINICAL TRIAL: NCT05298241
Title: Effects of Interactive Hand-grip Strength Game in Critically Illness Patients: A Randomized Controlled Trial
Brief Title: Interactive Hand-grip Strength Game in Critically Illness Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Associated professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202102007
Record Dates: First submitted 2022-01-30; First posted 2022-03-28 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Critical Illness
Keywords: intensive care unit; Hand-grip Strength
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand-grip Strength Game (Experimental): Participants will receive a hand-grip strength game for 5-20 minutes twice a day for consecutive three days.
  Interventions: Other: Hand-grip Strength Game
- routine care (No Intervention): The control group will not involve hand-grip strength game at night.

INTERVENTIONS:
Other: Hand-grip Strength Game — Interactive Handgrip Strength Game for ICU patients receiving the game and to assess the impact on psychological.
  Arms: Hand-grip Strength Game

SUMMARY:
Patients admitted to the intensive care units (ICUs) are an unexpected event that consequently causes physical and psychological problems, including ICU acquired weakness, delirium, sleep disruptions, anxiety, depression, and post-traumatic stress disorder (PTSD). Such consequences may lead to prolonged ICU stay, increased health care, and elevated medical costs. Therefore, mitigating physical and psychological distresses by providing timely effective interventions has become a top concern to optimize critically ill patients' recovery. Investigators aim to design an interactive hand-grip game to improve patients' upper limbs activities and psychological health in patients requiring intensive care.

DETAILED DESCRIPTION:
Patients admitted to the intensive care units (ICUs) are an unexpected event that consequently causes physical and psychological problems, including ICU acquired weakness, delirium, sleep disruptions, anxiety, depression, and post-traumatic stress disorder (PTSD). Such consequences may lead to prolonged ICU stay, increased health care, and elevated medical costs. Therefore, mitigating physical and psychological distresses by providing timely effective interventions has become a top concern to optimize critically ill patients' recovery. Investigaters aim to design a interactive hand-grip game to improve patients' upper limbs activities and psychological health in patients requiring intensive care. This will be a two-arm, parallel randomized controlled trial which randomly assign patients into the game group and usual care group.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 20 years
* Having clear consciousness
* Independently able to mobilize to complete the intervention and communicate in Chinese
* Richmond Agitation-Sedation Scale (RASS) 24 between +1 to -1 if using sedatives

Exclusion Criteria:

* Suspect neurological deficits
* Neuromuscular disease
* Orthopedic injuries with contraindications to mobilize

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline on anxiety | The 1 day of enrollment, and 3th day of ICU.
  Anxiety will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 of anxiety has 7 items of the questions are used to measure the severity of anxiety. The total score should be multiplied by 2 range from 0-42, if score>7 is associated with anxiety. The higher score means more severe anxiety.
Change from baseline on Post-traumatic stress disorder(PTSD) | The 1st, and 3th day of ICU.
  The PTSD is assessed by Post-traumatic Stress Syndrome 10-question inventory (PTSS-10).The measurement involved 10 items and each item is rated using a seven-point Likert scale (1 "never" to 7 "always").
Change of Delirium incidence | Every 8 hours during ICU stay up to 3 days
  The delirium event is assessed by Confusion Assessment Method for the ICU(CAM-ICU)
Change from baseline on depression | The 1 day of enrollment, and 3th day of ICU.
  Depression will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 7 items of the questions are used to measure the severity of depression. The total score should be multiplied by 2 range from 0-42, if score>9 is associated with depression. The higher score means more severe depression.
Change from baseline on stress | The 1 day of enrollment, and 3th day of ICU.
  Stress will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 7 items of the questions are used to measure the severity of stress. The total score should be multiplied by 2 range from 0-42, if score>14 is associated with anxiety. The higher score means more severe stress.

SECONDARY OUTCOMES:
Changes of Pain | Everyday during ICU stay up to 3 days
  Pain is assessed by using the Critical-Care Pain Observation Tool (CPOT). The possible total score ranges from 0 (no pain) to 8 (maximum pain).
Change from baseline on sleep quality | The 1st, and 3th day of ICU.
  Sleep quality in ICU is assessed by the Richards-Campbell Sleep Questionnaire(RCSQ). The mean of total score is 0-100. The higher score means the better sleep quality.
ICU acquired weakness | The 1st day of ICU.
  The ICU acquired weakness is assessed by Medical Research Council (MRC).The scale for grading the strength (i.e., 0, total palsy to 5, normal strength) in three functional muscle groups of each extremity (shoulder abduction, elbow flexion, and wrist extension for upper limb; hip flexion, knee extension, and ankle dorsiflexion for lower limb), with mean MRC-scores of <4 (antigravity strength).26,35 Summation of scores gives MRC-sums core, ranging from 0 to 60. The sum score also reliably identifies significant ICU-acquired weakness (< 48).

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Yean Chiu, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, Taipei, Taiwan